CLINICAL TRIAL: NCT06097273
Title: A Phase 3, Randomized, Observer-Blind, Active-Control Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1083 (SARS-CoV-2 and Influenza) Vaccine in Healthy Adult Participants, ≥50 Years of Age
Brief Title: A Study of mRNA-1083 (SARS-CoV-2 and Influenza) Vaccine in Healthy Adult Participants, ≥50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1083-P301
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2; Influenza
Keywords: mRNA-1083; mRNA-1083 Vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; Influenza Vaccine; Moderna
MeSH Terms: conditions — Influenza, Human; Coronavirus Infections; Virus Diseases | interventions — Influenza Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: mRNA-1083 and Placebo (Experimental): Participants of age 65 years and older will receive mRNA-1083 and placebo administered as 2 intramuscular (IM) injections of on Day 1.
  Interventions: Biological: mRNA-1083; Biological: Placebo
- Cohort A2: Influenza Vaccine and COVID-19 Vaccine (Active Comparator): Participants of age 65 years and older will receive age recommended quadrivalent influenza vaccine and COVID-19 vaccine administered as 2 IM injections on Day 1.
  Interventions: Biological: Influenza Vaccine; Biological: COVID-19 Vaccine
- Cohort B1: mRNA-1083 and Placebo (Experimental): Participants of age 50 to <65 years will receive mRNA-1083 and placebo administered as 2 IM injections of on Day 1.
  Interventions: Biological: mRNA-1083; Biological: Placebo
- Cohort B2: Influenza Vaccine and COVID-19 Vaccine (Active Comparator): Participants of age 50 to <65 years will receive age recommended quadrivalent influenza vaccine and COVID-19 vaccine administered as 2 IM injections on Day 1.
  Interventions: Biological: Influenza Vaccine; Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: mRNA-1083 — Suspension for injection
  Arms: Cohort A1: mRNA-1083 and Placebo; Cohort B1: mRNA-1083 and Placebo
Biological: Placebo — 0.9% sodium chloride suspension for injection
  Arms: Cohort A1: mRNA-1083 and Placebo; Cohort B1: mRNA-1083 and Placebo
Biological: Influenza Vaccine — Commercially available formulation (Suspension for injection [pre-filled syringe])
  Arms: Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Biological: COVID-19 Vaccine — Commercially available formulation (Suspension for injection)
  Arms: Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Cohort B2: Influenza Vaccine and COVID-19 Vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety, and reactogenicity of mRNA-1083 as compared with active control, co-administered licensed influenza and severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) vaccines, in 2 independent age-group sub-study cohorts, healthy adults 65 years and older (Cohort A) and healthy adults 50 to <65 years of age (Cohort B).

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy adults either ≥65 years of age (Cohort A) or 50 to <65 years of age (Cohort B) at the time of consent (Screening Visit).
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, and agreement to continue adequate contraception through 3 months following vaccine administration.
* Fully vaccinated for COVID-19 primary series according to the locally authorized or approved regimen, and their last COVID-19 vaccine (primary series or booster) was ≥90 days prior to Day 1.

Exclusion Criteria:

* Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants for >14 days in total within 180 days prior to Day 1 (for corticosteroids, ≥10 milligrams [mg]/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study. Inhaled nasal and topical steroids are allowed.
* Received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days prior to study injections or plans to receive a vaccine authorized or approved by a local health agency within 28 days after the study injections.
* Received a seasonal influenza vaccine ≤150 days prior to Day 1.
* Tested positive for influenza by local health authority-approved testing methods ≤150 days prior to Day 1.
* Has had close contact to someone with COVID-19 as defined by the Centers for Disease Control and Prevention (CDC) in the past 10 days prior to Day 1.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8061 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (145):
- United States (145):
  - Pinnacle Research Group-409 E 10th St, Anniston, Alabama
  - Accel Research Site - Achieve - Birmingham, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Desert Clinical Research - CCT - PPDS, Mesa, Arizona
  - Foothills Research Center - CCT - PPDS, Phoenix, Arizona
  - Headlands Research - Scottsdale - PPDS, Scottsdale, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Fiel Family & Sports Medicine - PC - CCT - PPDS, Tempe, Arizona
  - AES - DRS - Synexus Clinical Research US, Inc. - Cerritos, Cerritos, California
  - Long Beach Research Institute, LLC, Long Beach, California
  - CenExel Apex (CNS) - Los Alamitos - PPDS, Los Alamitos, California
  - Central Valley Research, LLC, Modesto, California
  - Carbon Health- NoHo West Urgent Care and Primary Care, North Hollywood, California
  - Empire Clinical Research, Pomona, California
  - Artemis Institute For Clinical Research LLC - Riverside - Headlands - PPDS, Riverside, California
  - Clinical Innovations Trials - Riverside - CenExel - PPDS, Riverside, California
  - Peninsula Research Associates - Headlands - PPDS, Rolling Hills Estates, California
  - Artemis Institute For Clinical Research LLC - San Diego - Headlands - PPDS, San Diego, California
  - AES - DRS - Synexus Clinical Research US, Inc. - Vista, Vista, California
  - Tekton Research - Fort Collins - PPDS, Fort Collins, Colorado
  - Tekton Research - Longmont - PPDS, Longmont, Colorado
  - Stamford Therapeutics Consortium - ERN - PPDS, Stamford, Connecticut
  - Chase Medical Research LLC - Waterbury, Waterbury, Connecticut
  - Revival Research Corporation, Doral, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - CenExel RCA - Hollywood, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Health Awareness - Jupiter - ERN - ERN, Jupiter, Florida
  - Accel Research Sites - Saint Petersburg - Largo - ERN - PPDS, Largo, Florida
  - Flourish Research - Leesburg - PPDS, Leesburg, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - AES - DRS - Optimal Research Florida - Melbourne, Melbourne, Florida
  - Suncoast Research Group LLC - Flourish - PPDS, Miami, Florida
  - St. Johns Center for Clinical Research - ERN - PPDS, Saint Augustine, Florida
  - ForCare Clinical Research - CenExel FCR - PPDS, Tampa, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - Atlanta, Atlanta, Georgia
  - DelRicht Research, LLC - Springer Wellness & Restorative - Atlanta - PPDS, Atlanta, Georgia
  - iResearch Atlanta - CenExel - PPDS, Decatur, Georgia
  - Javara, Inc./Privia Medical Group Georgia, LLC - Fayetteville - Javara - PPDS, Fayetteville, Georgia
  - Georgia Clinic - CCT - PPDS, Norcross, Georgia
  - Privia Medical Group Georgia, LLC - Savannah - Javara - PPDS, Savannah, Georgia
  - Clinical Research Atlanta - ERN - PPDS, Stockbridge, Georgia
  - AES - DRS - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - Cedar Crosse Research Center, Chicago, Illinois
  - Flourish Research - Andersonville - PPDS, Chicago, Illinois
  - Koch Family Medicine, Morton, Illinois
  - AES - DRS - Optimal Research Illinois - Peoria, Peoria, Illinois
  - DM Clinical Research - Chicago - ERN - PPDS, River Forest, Illinois
  - AES - DRS - Synexus Clinical Research US, Inc. - Evansville, Evansville, Indiana
  - Velocity Clinical Research - Valparaiso (Buynak Clinical Research) - PPDS, Valparaiso, Indiana
  - The Iowa Clinic, P.C. - West Des Moines Campus, West Des Moines, Iowa
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Delricht Overland Park, Overland Park, Kansas
  - Tekton Research - Wichita - PPDS, Wichita, Kansas
  - DelRicht Research, LLC - Louisville - PPDS, Louisville, Kentucky
  - Versailles Family Medicine - CCT - PPDS, Versailles, Kentucky
  - Velocity Clinical Research (Baton Rouge - Louisiana) - PPDS, Baton Rouge, Louisiana
  - Velocity Clinical Research - Covington - PPDS, Covington, Louisiana
  - DelRicht Clinical Research, LLC - The Murphy Clinic - PPDS, Mandeville, Louisiana
  - IMA Clinical Research - Monroe, LA - PPDS, Monroe, Louisiana
  - DelRicht Clinical Research, LLC - New Orleans - ClinEdge - PPDS, New Orleans, Louisiana
  - DelRicht Research, LLC - Internal - Baton Rouge - PPDS, Prairieville, Louisiana
  - Annapolis Internal Medicine - CCT - PPDS, Annapolis, Maryland
  - Advanced Primary Care & Geriatric Care - CCT - PPDS, Rockville, Maryland
  - DelRicht Clinical Research, LLC - Matthew Mintz, MD - PPDS, Rockville, Maryland
  - Velocity Clinical Research (Rockville - Maryland) - PPDS, Rockville, Maryland
  - Privia Medical Group, LLC - Columbia Pike - Silver Spring - Javara - PPDS, Silver Spring, Maryland
  - DM Clinical Research - The Brook House - ERN - PPDS, Brookline, Massachusetts
  - Headlands Research - Detroit - Headlands - PPDS, Southfield, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research - Southfield - ERN - PPDS, Southfield, Michigan
  - Mankato Clinic - Premier Drive - Javara - PPDS, Mankato, Minnesota
  - AES - DRS - Synexus Clinical Research US, Inc. - Minneapolis, Richfield, Minnesota
  - DelRicht Research, LLC - Gulfport - PPDS, Gulfport, Mississippi
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Louis, Creve Coeur, Missouri
  - Clay Platte Family Medicine - CCT Research, Kansas City, Missouri
  - Clinvest - National Ave - Headlands - PPDS, Springfield, Missouri
  - DelRicht Research, LLC - Command Family Medicine - Springfield - DelRicht - PPDS, Springfield, Missouri
  - Sundance Clinical Research - ERN - PPDS, St Louis, Missouri
  - DelRicht Clinical Research, LLC - MS. Medicine - PPDS, Town and Country, Missouri
  - Skyline Medical Center - PC - CCT - PPDS, Elkhorn, Nebraska
  - Methodist Physicians Clinic - CCT Research - PPDS, Fremont, Nebraska
  - Velocity Clinical Research (Lincoln - Nebraska) - PPDS, Lincoln, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Midwest Regional Health Services - LLC - CCT - PPDS, Omaha, Nebraska
  - Papillion Research Center, Papillion, Nebraska
  - AES - DRS - Synexus Clinical Research US, Inc. - Henderson, Henderson, Nevada
  - Santa Rosa Urgent Care - Primary Care - CCT - PPDS, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Hassman Research Institute - HRI - Berlin - CenExel - PPDS, Berlin, New Jersey
  - Velocity Clinical Research - Albuquerque - PPDS, Albuquerque, New Mexico
  - AXCES Research Group - Sante Fe - ERN - PPDS, Santa Fe, New Mexico
  - DM Clinical Research - Brooklyn, Brooklyn, New York
  - AES - DRS - Synexus Clinical Research US, Inc. - New York, New York, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - DelRicht Research, LLC - Charlotte - PPDS, Charlotte, North Carolina
  - Tryon Medical Partners, PLLC and Javara Inc. - Javara - PPDS, Charlotte, North Carolina
  - Monroe Biomedical Research -343 Venus St, Monroe, North Carolina
  - Trial Management Associates LLC - ERN - PPDS, Wilmington, North Carolina
  - CTI Clinical Research Center - PPDS, Cincinnati, Ohio
  - Velocity Clinical Research (Cincinnati - Ohio) - PPDS, Cincinnati, Ohio
  - AES - DRS - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - AES - DRS - Synexus Clinical Research US, Inc. - Columbus, Columbus, Ohio
  - WellNow Urgent Care & Research - Huber Heights, Huber Heights, Ohio
  - Tekton Research - Edmond - PPDS, Edmond, Oklahoma
  - Lynn Institute of East Oklahoma - ERN - PPDS, Oklahoma City, Oklahoma
  - DelRicht Research, LLC - Internal - Tulsa - PPDS, Tulsa, Oklahoma
  - Tekton Research - Yukon - PPDS, Yukon, Oklahoma
  - The Corvallis Clinic, PC - 3680 NW Samaritan Drive, Corvallis, Oregon
  - Hatboro Medical Associates - CCT - PPDS, Hatboro, Pennsylvania
  - DM Clinical Research - Philadelphia - ERN - PPDS, Philadelphia, Pennsylvania
  - AES - DRS - Synexus Clinical Research US, Inc. - Anderson, Anderson, South Carolina
  - TMA - Myrtle Beach - ERN - PPDS, Myrtle Beach, South Carolina
  - Velocity Clinical Research - Spartanburg - PPDS, Spartanburg, South Carolina
  - DelRicht Research, LLC - Hendersonville - PPDS, Hendersonville, Tennessee
  - AES - DRS - Optimal Research Texas - Austin, Austin, Texas
  - Benchmark Research - Austin - HyperCore - PPDS, Austin, Texas
  - Tekton Research - Austin - PPDS, Austin, Texas
  - Tekton Research Inc, Beaumont, Texas
  - Headlands Research - Brownsville - Headlands - PPDS, Brownsville, Texas
  - AES - DRS - Synexus Clinical Research US, Inc. - Dallas, Dallas, Texas
  - 3A Research, LLC, El Paso, Texas
  - Privia Medical Group- North Texas - West Parker Road - Fort Worth - Javara - PPDS, Fort Worth, Texas
  - Mount Olympus Medical Research Group - ClinEdge - PPDS, Friendswood, Texas
  - DM Clinical Research - Cyfair Clinical Research Center - ERN - PPDS, Houston, Texas
  - DM Clinical Research - Bellaire - ERN - PPDS, Houston, Texas
  - DM Clinical Research - Texas Center for Drug Development - Humble - ERN - PPDS, Humble, Texas
  - DelRicht Research, LLC - Zomnir Family Medicine - DelRicht - PPDS, McKinney, Texas
  - Benchmark Research - San Angelo - HyperCore - PPDS, San Angelo, Texas
  - Sun Research Institute -427 9th St, San Antonio, Texas
  - Clinical Trials of Texas, Inc. - PPDS, San Antonio, Texas
  - IMA Clinical Research - San Antonio - PPDS, San Antonio, Texas
  - Tekton Research - San Antonio - PPDS, San Antonio, Texas
  - Privia Medical Group Gulf Coast, PLLC - San Marcos - Javara - PPDS, San Marcos, Texas
  - Privia Medical Group- North Texas - Stephenville - Javara - PPDS, Stephenville, Texas
  - DM Clinical Research - Sugarland - ERN - PPDS, Sugar Land, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - Cope Family Medicine - CCT - PPDS, Bountiful, Utah
  - Ogden Clinic - Mountain View - CCT - PPDS, Pleasant View, Utah
  - Ogden Clinic - Grandview - CCT - PPDS, Roy, Utah
  - JBR Clinical Research - CenExel JBR - PPDS, Salt Lake City, Utah
  - AES - DRS - Synexus Clinical Research US, Inc. - Salt Lake City, South Salt Lake, Utah
  - Velocity Clinical Research - Family Practice - Portsmouth - PPDS, Portsmouth, Virginia
  - Wenatchee Valley Hospital & Clinics Campus, Wenatchee, Washington

REFERENCES:
- [Derived] Rudman Spergel AK, Wu I, Deng W, Cardona J, Johnson K, Espinosa-Fernandez I, Sinkiewicz M, Urdaneta V, Carmona L, Schaefers K, Girard B, Paila YD, Mehta D, Callendret B, Kostanyan L, Ananworanich J, Miller J, Das R, Shaw CA. Immunogenicity and Safety of Influenza and COVID-19 Multicomponent Vaccine in Adults >/=50 Years: A Randomized Clinical Trial. JAMA. 2025 Jun 10;333(22):1977-1987. doi: 10.1001/jama.2025.5646. PMID 40332892
- [Derived] Sanchez-Martinez ZV, Alpuche-Lazcano SP, Stuible M, Akache B, Renner TM, Deschatelets L, Dudani R, Harrison BA, McCluskie MJ, Hrapovic S, Blouin J, Wang X, Schuller M, Cui K, Cho JY, Durocher Y. SARS-CoV-2 spike-based virus-like particles incorporate influenza H1/N1 antigens and induce dual immunity in mice. Vaccine. 2024 Dec 2;42(26):126463. doi: 10.1016/j.vaccine.2024.126463. Epub 2024 Oct 30. PMID 39481241

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A1: mRNA-1083 and Placebo: Participants of age 65 years and older received mRNA-1083 and placebo administered as 2 intramuscular (IM) injections (1 in each deltoid muscle) on Day 1.
- Cohort A2: Influenza Vaccine and COVID-19 Vaccine: Participants of age 65 years and older received age recommended influenza vaccine and coronavirus disease 2019 (COVID-19) vaccine administered as 2 IM injections (1 in each deltoid muscle) on Day 1.
- Cohort B1: mRNA-1083 and Placebo: Participants of age 50 to <65 years received mRNA-1083 and placebo administered as 2 IM injections (1 in each deltoid muscle) on Day 1.
- Cohort B2: Influenza Vaccine and COVID-19 Vaccine: Participants of age 50 to <65 years received age recommended influenza vaccine and COVID-19 vaccine administered as 2 IM injections (1 in each deltoid muscle) on Day 1.
Period: Overall Study
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Started | 2025 | 2012 | 2009 | 2015
Received Both Injections | 2011 | 2006 | 1993 | 2005
Completed | 1974 | 1977 | 1944 | 1957
Not Completed | 51 | 35 | 65 | 58
Not completed — Death | 2 | 1 | 2 | 2
Not completed — Lost to Follow-up | 27 | 18 | 36 | 31
Not completed — Physician Decision | 0 | 1 | 0 | 3
Not completed — Protocol Violation | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 11 | 14 | 15
Not completed — Other Than Specified | 7 | 3 | 11 | 6

BASELINE CHARACTERISTICS:
Population: The randomization set included all participants who were randomly assigned. Participants were included in the treatment arm to which they were randomized.
Groups:
- Cohort A1: mRNA-1083 and Placebo: Participants of age 65 years and older received mRNA-1083 and placebo administered as 2 IM injections (1 in each deltoid muscle) on Day 1.
- Cohort A2: Influenza Vaccine and COVID-19 Vaccine: Participants of age 65 years and older received age recommended influenza vaccine and COVID-19 vaccine administered as 2 IM injections (1 in each deltoid muscle) on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine | Total
Number analyzed (Participants) | 2025 | 2012 | 2009 | 2015 | 8061
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (4.96) | 70.7 (4.70) | 57.5 (4.25) | 57.4 (4.21) | 64.1 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1084 | 1100 | 1165 | 1201 | 4550
  Male | 941 | 912 | 844 | 814 | 3511
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 284 | 275 | 393 | 381 | 1333
  Not Hispanic or Latino | 1701 | 1695 | 1591 | 1613 | 6600
  Unknown or Not Reported | 40 | 42 | 25 | 21 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1588 | 1570 | 1382 | 1350 | 5890
  Race: Black or African American | 373 | 370 | 522 | 555 | 1820
  Race: Asian | 25 | 37 | 52 | 39 | 153
  Race: American Indian or Alaska Native | 9 | 12 | 12 | 13 | 46
  Race: Native Hawaiian or Other Pacific Islander | 1 | 4 | 3 | 5 | 13
  Race: Other | 4 | 3 | 4 | 8 | 19
  Race: Multiple | 14 | 4 | 19 | 21 | 58
  Race: Unknown/Not Reported | 11 | 12 | 15 | 24 | 62

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean (GM) Level of Antibodies for Influenza, as Measured by Hemagglutination Inhibition (HAI) Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. The Per Protocol Immunogenicity Set (PPIS) included all randomized participants who received study intervention, complied with the timing of immunogenicity blood sample collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative reverse transcription polymerase chain reaction (RT-PCR) test for influenza and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Day 29
Population: The PPIS. Overall number of participants analyzed = participants evaluable for this outcome measure. Number Analyzed = participants evaluable for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 1885 | 1883 | 1889 | 1883
titer
  Influenza A H1N1 Antibody | 120.5 [116.0 to 125.2] | 104.3 [100.4 to 108.4] | 137.7 [132.1 to 143.5] | 97.3 [93.4 to 101.5]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 1885 | 1883 | 1889 | 1882
  Influenza A H3N2 Antibody | 114.7 [110.4 to 119.2] | 107.9 [103.9 to 112.1] | 111.5 [107.5 to 115.7] | 80.8 [77.9 to 83.8]
  Influenza B Victoria-lineage Antibody | 245.3 [237.8 to 252.9] | 219.4 [212.8 to 226.3] | 224.9 [218.0 to 232.0] | 185.0 [179.3 to 190.8]
  Influenza B Yamagata-lineage Antibody: number analyzed (Participants) | 1885 | 1883 | 1889 | 1882
  Influenza B Yamagata-lineage Antibody | 93.3 [91.1 to 95.6] | 92.6 [90.4 to 94.9] | 101.7 [99.3 to 104.3] | 88.1 [86.0 to 90.3]
Statistical Analysis 1: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza A H1N1 Antibody; Test type: Non-Inferiority — The noninferiority in GM level in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 97.5% CI of the GMR was >0.667; GMR = 1.155, 97.5% CI 2-sided [1.086 to 1.229]
Statistical Analysis 2: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza A H1N1 Antibody; Test type: Superiority — The superiority in GM level in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 95% confidence interval (CI) of the geometric mean ratio (GMR) was >1; GMR = 1.155, 95% CI 2-sided [1.094 to 1.220]
Statistical Analysis 3: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza A H3N2 Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR = 1.063, 97.5% CI 2-sided [0.999 to 1.130]
Statistical Analysis 4: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza A H3N2 Antibody; Test type: Superiority — The superiority in GM level in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 95% CI of the GMR was >1; GMR = 1.063, 95% CI 2-sided [1.007 to 1.122]
Statistical Analysis 5: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza A H1N1 Antibody; Test type: Non-Inferiority — The noninferiority in GM level in the Cohort B1 group compared with that of Cohort B2 group was demonstrated if the lower bound of the 97.5% CI of the GMR was >0.667; GMR = 1.414, 97.5% CI 2-sided [1.322 to 1.513]
Statistical Analysis 6: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza A H1N1 Antibody; Test type: Superiority — The superiority in GM level in the Cohort B1 group compared with that of Cohort B2 group was demonstrated if the lower bound of the 95% CI of the GMR was >1; GMR = 1.414, 95% CI 2-sided [1.333 to 1.500]
Statistical Analysis 7: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza A H3N2 Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 5]; GMR = 1.380, 97.5% CI 2-sided [1.300 to 1.465]
Statistical Analysis 8: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza A H3N2 Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 6]; GMR = 1.380, 95% CI 2-sided [1.310 to 1.454]
Statistical Analysis 9: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza B Victoria-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR = 1.118, 97.5% CI 2-sided [1.063 to 1.175]
Statistical Analysis 10: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza B Victoria-lineage Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 4]; GMR = 1.118, 95% CI 2-sided [1.070 to 1.167]
Statistical Analysis 11: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza B Yamagata-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR = 1.007, 97.5% CI 2-sided [0.969 to 1.047]
Statistical Analysis 12: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for Influenza B Yamagata-lineage Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 4]; GMR = 1.007, 95% CI 2-sided [0.973 to 1.042]
Statistical Analysis 13: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza B Victoria-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 5]; GMR = 1.216, 97.5% CI 2-sided [1.156 to 1.278]
Statistical Analysis 14: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza B Victoria-lineage Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 6]; GMR = 1.216, 95% CI 2-sided [1.163 to 1.270]
Statistical Analysis 15: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza B Yamagata-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 5]; GMR = 1.154, 97.5% CI 2-sided [1.109 to 1.201]
Statistical Analysis 16: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for Influenza B Yamagata-lineage Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 6]; GMR = 1.154, 95% CI 2-sided [1.115 to 1.195]

2. Primary Outcome: GM Level of Antibodies for SARS-CoV-2, as Measured by Pseudovirus Neutralization Assay (PsVNA)
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. The PPIS included all randomized participants who received study intervention, complied with the timing of immunogenicity blood sample collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Day 29
Population: The PPIS. Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 1849 | 1859 | 1854 | 1848
titer | 1396.7 [1326.6 to 1470.5] | 851.1 [808.6 to 895.9] | 1551.6 [1476.3 to 1630.7] | 1186.1 [1128.5 to 1246.7]
Statistical Analysis 1: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for SARS-CoV-2 Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 4]; GMR = 1.641, 95% CI 2-sided [1.526 to 1.765]
Statistical Analysis 2: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort A1 vs Cohort A2) for SARS-CoV-2 Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR = 1.641, 97.5% CI 2-sided [1.510 to 1.783]
Statistical Analysis 3: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for SARS-CoV-2 Antibody; Test type: Superiority — [test comment as in outcome 1, analysis 6]; GMR = 1.308, 95% CI 2-sided [1.219 to 1.404]
Statistical Analysis 4: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; GMR (Cohort B1 vs Cohort B2) for SARS-CoV-2 Antibody; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 5]; GMR = 1.308, 97.5% CI 2-sided [1.207 to 1.418]

3. Primary Outcome: Influenza: Percentage of Participants With Seroconversion, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Seroconversion was defined as a Day 29 postinjection level ≥1:40 if Baseline was <1:10 or a 4-fold or greater rise if Baseline was ≥1:10 in anti-hemagglutinin (HA) antibodies measured by HAI assay. The PPIS included all randomized participants who received study intervention, complied with the timing of immunogenicity blood sample collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 1885 | 1883 | 1888 | 1882
percentage of participants
  Influenza A H1N1 Antibody | 36.4 [34.3 to 38.7] | 31.1 [29.0 to 33.2] | 50.6 [48.3 to 52.9] | 32.7 [30.6 to 34.8]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 1885 | 1883 | 1888 | 1881
  Influenza A H3N2 Antibody | 38.7 [36.5 to 40.9] | 34.6 [32.5 to 36.8] | 41.9 [39.7 to 44.2] | 27.4 [25.4 to 29.5]
  Influenza B Victoria-lineage Antibody | 23.9 [22.0 to 25.9] | 19.4 [17.6 to 21.2] | 25.8 [23.9 to 27.9] | 17.2 [15.5 to 19.0]
  Influenza B Yamagata-lineage Antibody: number analyzed (Participants) | 1885 | 1883 | 1888 | 1881
  Influenza B Yamagata-lineage Antibody | 8.8 [7.5 to 10.1] | 10.2 [8.9 to 11.7] | 13.0 [11.5 to 14.6] | 10.3 [9.0 to 11.8]
Statistical Analysis 1: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Influenza A H1N1 Antibody; Test type: Superiority — The superiority in seroconversion rate (SCR) in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 95% CI of the SCR difference was >0%; Percentage Difference = 5.4, 95% CI 2-sided [2.4 to 8.4]
Statistical Analysis 2: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Influenza A H1N1 Antibody; Test type: Non-Inferiority — The noninferiority in SCR in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 97.5% CI of the SCR difference was >-10%; Percentage Difference = 5.4, 97.5% CI 2-sided [1.9 to 8.8]
Statistical Analysis 3: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Influenza A H3N2 Antibody; Test type: Superiority — The superiority in SCR in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 95% CI of the SCR difference was >0%; Percentage Difference = 4.0, 95% CI 2-sided [1.0 to 7.1]
Statistical Analysis 4: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Influenza A H3N2 Antibody; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Percentage Difference = 4.0, 97.5% CI 2-sided [0.5 to 7.6]
Statistical Analysis 5: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Victoria-lineage Antibody; Test type: Superiority — [test comment as in outcome 3, analysis 3]; Percentage Difference = 4.5, 95% CI 2-sided [1.9 to 7.2]
Statistical Analysis 6: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Victoria-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Percentage Difference = 4.5, 95% CI 2-sided [1.5 to 7.5]
Statistical Analysis 7: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Yamagata-lineage Antibody; Test type: Superiority — [test comment as in outcome 3, analysis 3]; Percentage Difference = -1.4, 95% CI 2-sided [-3.3 to 0.4]
Statistical Analysis 8: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for Yamagata-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Percentage Difference = -1.4, 97.5% CI 2-sided [-3.6 to 0.7]
Statistical Analysis 9: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Influenza A H1N1 Antibody; Test type: Superiority — The superiority in SCR in the Cohort B1 group compared with that of Cohort B2 group was demonstrated if the lower bound of the 95% CI of the SCR difference was >0%; Percentage Difference = 17.9, 95% CI 2-sided [14.8 to 21.0]
Statistical Analysis 10: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Influenza A H1N1 Antibody; Test type: Non-Inferiority — The noninferiority in SCR in the Cohort B1 group compared with that of Cohort B2 group was demonstrated if the lower bound of the 97.5% CI of the SCR difference was >-10%; Percentage Difference = 17.9, 97.5% CI 2-sided [14.3 to 21.4]
Statistical Analysis 11: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Influenza A H3N2 Antibody; Test type: Superiority — [test comment as in outcome 3, analysis 9]; Percentage Difference = 14.6, 95% CI 2-sided [11.6 to 17.6]
Statistical Analysis 12: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Influenza A H3N2 Antibody; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Percentage Difference = 14.6, 97.5% CI 2-sided [11.1 to 18.0]
Statistical Analysis 13: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Victoria-lineage Antibody; Test type: Superiority — [test comment as in outcome 3, analysis 9]; Percentage Difference = 8.6, 95% CI 2-sided [6.0 to 11.2]
Statistical Analysis 14: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Victoria-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Percentage Difference = 8.6, 97.5% CI 2-sided [5.6 to 11.6]
Statistical Analysis 15: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Yamagata-lineage Antibody; Test type: Superiority — [test comment as in outcome 3, analysis 9]; Percentage Difference = 2.7, 95% CI 2-sided [0.6 to 4.7]
Statistical Analysis 16: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for Yamagata-lineage Antibody; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 10]; Percentage Difference = 2.7, 97.5% CI 2-sided [0.3 to 5.0]

4. Primary Outcome: SARS-CoV-2: Percentage of Participants With Seroresponse, as Measured by PsVNA
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Seroresponse was defined as a Day 29 postinjection level ≥4-fold rise if Baseline was ≥lower limit of quantification (LLOQ) or ≥4×LLOQ if Baseline value was <LLOQ in the nAb values measured by PsVNA. LLOQ was 38 arbitrary unit (AU)/milliliter (mL). The PPIS included all randomized participants who received study intervention, complied with the timing of immunogenicity blood sample collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Baseline to Day 29
Population: The PPIS. Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 1841 | 1854 | 1852 | 1846
percentage of participants | 82.3 [80.5 to 84.1] | 69.6 [67.4 to 71.7] | 84.6 [82.8 to 86.2] | 76.5 [74.5 to 78.4]
Statistical Analysis 1: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for SARS-CoV-2 Antibody; Test type: Superiority — The superiority in seroresponse rate (SRR) in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 95% CI of the SRR difference was >0%; Percentage Difference = 12.8, 95% CI 2-sided [10.0 to 15.5]
Statistical Analysis 2: Comparison: Cohort A1: mRNA-1083 and Placebo vs Cohort A2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort A1 vs Cohort A2) for SARS-CoV-2 Antibody; Test type: Non-Inferiority — The noninferiority in SRR in the Cohort A1 group compared with that of Cohort A2 group was demonstrated if the lower bound of the 97.5% CI of the SRR difference was >-10%; Percentage Difference = 12.8, 97.5% CI 2-sided [9.6 to 15.9]
Statistical Analysis 3: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for SARS-CoV-2 Antibody; Test type: Superiority — The superiority in SRR in the Cohort B1 group compared with that of Cohort B2 group was demonstrated if the lower bound of the 95% CI of the SRR difference was >0%; Percentage Difference = 8.1, 95% CI 2-sided [5.5 to 10.6]
Statistical Analysis 4: Comparison: Cohort B1: mRNA-1083 and Placebo vs Cohort B2: Influenza Vaccine and COVID-19 Vaccine; Percentage Difference (Cohort B1 vs Cohort B2) for SARS-CoV-2 Antibody; Test type: Non-Inferiority — The noninferiority in SRR in the Cohort B1 group compared with that of Cohort B2 group was demonstrated if the lower bound of the 97.5% CI of the SRR difference was >-10%; Percentage Difference = 8.1, 97.5% CI 2-sided [5.2 to 11.0]

5. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were reported by participants an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. All solicited ARs considered causally related to injection were graded 0-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicates lower severity, and a higher score indicates greater severity. The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Up to 7 days after study injection
Population: The Solicited Safety Set included all randomized participants who received any study vaccination and contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 2011 | 2001 | 1993 | 2004
Participants
  Any | 1681 | 1565 | 1698 | 1640
  Grade 3 or Grade 4 | 183 | 84 | 246 | 127

6. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Number of participants with unsolicited AEs (SAEs and non-serious AEs) up to 28 days post-vaccination are reported in this outcome measure. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Up to 28 days after study injection
Population: The Safety Set included all participants who were randomized and received any study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 2011 | 2006 | 1993 | 2005
Participants | 239 | 250 | 195 | 191

7. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that lead to an unscheduled visit to an healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or COVID-19 and visits to healthcare practitioners external to the study site. Number of participants with SAEs, AESIs, MAAEs, and AEs leading to discontinuation up to the end of study (Day 181) are reported in this outcome measure. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 181
Population: The Safety Set included all participants who were randomized and received any study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 2011 | 2006 | 1993 | 2005
Participants
  SAEs | 70 | 52 | 29 | 27
  AESIs | 18 | 13 | 4 | 9
  MAAEs | 426 | 428 | 301 | 304
  AEs Leading to Discontinuation | 0 | 0 | 1 | 0

8. Secondary Outcome: Geometric Mean Fold-Rise (GMFR) of Antibodies for Influenza, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% CI for GMFR was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation. PPIS included all randomized participants who received study intervention, complied with the timing of immunogenicity blood sample collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Day 1, Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 1885 | 1883 | 1888 | 1882
ratio
  Influenza A H1N1 Antibody | 2.70 [2.60 to 2.81] | 2.36 [2.26 to 2.46] | 3.70 [3.54 to 3.86] | 2.54 [2.43 to 2.66]
  Influenza A H3N2 Antibody: number analyzed (Participants) | 1885 | 1883 | 1888 | 1881
  Influenza A H3N2 Antibody | 2.78 [2.67 to 2.89] | 2.59 [2.48 to 2.70] | 3.07 [2.95 to 3.19] | 2.22 [2.13 to 2.31]
  Influenza B Victoria-lineage | 2.05 [1.98 to 2.12] | 1.84 [1.77 to 1.90] | 2.13 [2.06 to 2.20] | 1.75 [1.69 to 1.81]
  Influenza B Yamagata-lineage: number analyzed (Participants) | 1885 | 1883 | 1888 | 1881
  Influenza B Yamagata-lineage | 1.52 [1.48 to 1.55] | 1.52 [1.48 to 1.56] | 1.71 [1.66 to 1.75] | 1.48 [1.44 to 1.52]

9. Secondary Outcome: GMFR of Antibodies for SARS-CoV-2, as Measured by PsVNA
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% CI for GMFR was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation. PPIS included all randomized participants who received study intervention, complied with the timing of immunogenicity blood sample collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Day 1, Day 29
Population: The PPIS. Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 1841 | 1854 | 1852 | 1846
ratio | 16.86 [15.87 to 17.93] | 10.32 [9.72 to 10.96] | 17.83 [16.78 to 18.94] | 13.56 [12.72 to 14.46]

10. Secondary Outcome: GM Level of Antibodies for Influenza, as Measured by Microneutralization (MN) Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. The PPIS for MN assay included a subset of randomized participants who received study intervention to be tested for MN, complied with the timing of immunogenicity blood sampling collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Day 29
Population: The PPIS for MN assay.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 146 | 146 | 147 | 147
titer
  Influenza A H1N1 Antibody | 676.4 [528.8 to 865.3] | 635.9 [489.4 to 826.4] | 946.8 [729.7 to 1228.4] | 428.1 [327.0 to 560.4]
  Influenza A H3N2 Antibody | 587.6 [483.9 to 713.6] | 668.8 [538.9 to 830.0] | 645.8 [519.1 to 803.5] | 393.9 [324.7 to 477.9]
  Influenza B Victoria-lineage Antibody | 2845.4 [2406.1 to 3364.9] | 3072.5 [2571.0 to 3671.9] | 2901.5 [2457.6 to 3425.6] | 1883.1 [1571.4 to 2256.5]
  Influenza B Yamagata-lineage Antibody | 1118.8 [910.4 to 1374.9] | 1434.4 [1200.9 to 1713.3] | 1449.6 [1222.5 to 1719.0] | 1071.3 [883.8 to 1298.4]

11. Secondary Outcome: GMFR of Antibodies for Influenza, as Measured by MN Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% CI for GMFR was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation. The PPIS for MN assay included a subset of randomized participants who received study intervention to be tested for MN, complied with the timing of immunogenicity blood sampling collections to have both Baseline and Day 29 assessments using a window of -7 to +14 days, had no major dosing error, had negative RT-PCR test for influenza and SARS-CoV-2 on Day 1, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Day 1, Day 29
Population: The PPIS for MN assay.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 146 | 146 | 147 | 147
ratio
  Influenza A H1N1 Antibody | 4.89 [3.92 to 6.10] | 4.68 [3.68 to 5.94] | 8.74 [7.03 to 10.87] | 5.14 [4.01 to 6.60]
  Influenza A H3N2 Antibody | 2.88 [2.44 to 3.41] | 2.46 [2.01 to 3.01] | 3.33 [2.76 to 4.01] | 1.94 [1.64 to 2.31]
  Influenza B Victoria-lineage | 3.22 [2.63 to 3.94] | 3.02 [2.48 to 3.67] | 3.87 [3.27 to 4.58] | 3.27 [2.66 to 4.02]
  Influenza B Yamagata-lineage | 2.98 [2.56 to 3.46] | 3.38 [2.75 to 4.15] | 3.66 [3.02 to 4.44] | 3.42 [2.79 to 4.19]

12. Other Pre Specified Outcome: Number of Deaths Related to Study Drug mRNA-1083 and Placebo
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, irrespective of its perceived relationship to the study drug. The Investigator assessed the causality by determining whether there was a reasonable possibility that the death was related to the study drug, using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable AND/OR the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable.
Time Frame: Day 1 through Day 181
Population: Safety set included all participants who were randomized and received any study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort B1: mRNA-1083 and Placebo
Number analyzed (Participants) | 2025 | 2009
Participants
  Deaths | 2 | 2
  Deaths Related to Study Drug mRNA-1083 | 0 | 0

13. Other Pre Specified Outcome: Number of Deaths Related to Control Drug Influenza Vaccine and COVID-19 Vaccine
Description: as for outcome 12
Time Frame: Day 1 through Day 181
Population: Safety set included all participants who were randomized and received any study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
Number analyzed (Participants) | 2012 | 2015
Participants
  Deaths | 1 | 2
  Deaths Related to Control Drug | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 181
Description: The all-cause mortality was based on the randomization set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all participants who were randomized and received any study vaccination.
Arm/Group | Cohort A1: mRNA-1083 and Placebo | Cohort A2: Influenza Vaccine and COVID-19 Vaccine | Cohort B1: mRNA-1083 and Placebo | Cohort B2: Influenza Vaccine and COVID-19 Vaccine
All-Cause Mortality (participants affected / at risk) | 2/2025 | 1/2012 | 2/2009 | 2/2015
Serious Adverse Events (participants affected / at risk) | 71/2011 | 52/2006 | 29/1993 | 27/2005
Other Adverse Events (participants affected / at risk) | 0/2011 | 0/2006 | 0/1993 | 0/2005
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: mRNA-1083 and Placebo (N=2011) | Cohort A2: Influenza Vaccine and COVID-19 Vaccine (N=2006) | Cohort B1: mRNA-1083 and Placebo (N=1993) | Cohort B2: Influenza Vaccine and COVID-19 Vaccine (N=2005)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Janus kinase 2 mutation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The Investigator considered this event related to mRNA-1083 investigational vaccine, while the Sponsor attributed it to pre-existing conditions and not related to mRNA-1083 investigational vaccine.
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The Investigator considered this event related to mRNA-1083 investigational vaccine, while the Sponsor attributed it to pre-existing conditions and not related to mRNA-1083 investigational vaccine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT06097273/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT06097273/SAP_001.pdf